CLINICAL TRIAL: NCT03520959
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Determine the Efficacy and Safety of CMB305 in Unresectable Locally-advanced or Metastatic NY-ESO-1+ Synovial Sarcoma Participants Following First Line Systemic Anti-cancer Therapy (V943-003, IMDZ-04-1702)
Brief Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study For Subjects With Locally-advanced Unresectable or Metastatic Synovial Sarcoma (V943-003, IMDZ-04-1702)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to sponsor's decision.
Sponsor: Immune Design, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMDZ-04-1702; V943A-003 (Other: Merck Unique ID)
Record Dates: First submitted 2018-03-30; First posted 2018-05-11 (Actual); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Synovial Sarcoma; Cancer; Soft Tissue Sarcoma; Sarcoma; Metastatic Sarcoma
Keywords: Synovate Study; NY-ESO-1; cancer vaccine; Sarcoma; soft tissue sarcoma; immunotherapy
MeSH Terms: conditions — Sarcoma, Synovial; Neoplasms; Sarcoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): A sequential regimen of LV305-matching placebo and G305-matching placebo.
  Interventions: Other: LV305-matching placebo; Other: G305-matching placebo
- CMB305 (Experimental): A sequential regimen of LV305 and G305.
  Interventions: Biological: LV305; Biological: G305

INTERVENTIONS:
Biological: LV305 — Administered via subcutaneous (SC) injection.
  Arms: CMB305
Biological: G305 — Administered via intramuscular (IM) injection.
  Arms: CMB305
Other: LV305-matching placebo — Administered via SC injection.
  Arms: Placebo
Other: G305-matching placebo — Administered via IM injection.
  Arms: Placebo

SUMMARY:
To assess if the CMB305 vaccine regimen may help the body's immune system to slow or stop the growth of synovial sarcoma tumor and improve survival.

DETAILED DESCRIPTION:
The Synovate Study is a global, randomized, double-blind, placebo-controlled, phase 3 study in patients with unresectable, locally-advanced or metastatic New York esophageal squamous cell carcinoma 1 (NY-ESO-1) positive synovial sarcoma following first-line systemic anti-cancer therapy.

ELIGIBILITY:
Selected Inclusion Criteria:

* Histological diagnosis of synovial sarcoma
* Immunohistochemistry (IHC) results from tumor biopsy for New York esophageal squamous cell carcinoma 1 (NY-ESO-1) are positive
* Participants have received at least 4 but no more than 8 cycles of first-line anthracycline or ifosfamide-containing systemic anti-cancer therapy regimen
* Must have documentation of no evidence of disease progression of the tumor during or after completion of first line systemic anti-cancer therapy
* ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1
* Age >/= 12 years
* Life expectancy of at least 6 months

Selected Exclusion Criteria:

* Have received last dose of first-line systemic anti-cancer therapy or date of most recent local regional therapy >28 days prior to day 1
* Have received prior anti-NY-ESO-1 therapy
* Have received first-line systemic anti-cancer therapy with an agent other than anthracycline or ifosfamide
* Have received treatment with systemic immunomodulatory agents within 28 days prior to administration of the first dose of CMB305, or 5 half-lives of the drug, whichever occurs sooner.
* Have significant immunosuppression from concurrent, recent, or anticipated need for chronic treatment with systemic immunosuppressive dose of corticosteroids or immunosuppressive medications.
* Have psychiatric or other medical illness, or any other condition that in the opinion of the investigator prevents compliance with the study procedures or ability to provide valid informed consent.
* Have history of uncontrolled autoimmune disease.
* Have a significant electrocardiogram finding or cardiovascular disease
* have inadequate organ function per protocol
* History of other cancer within 3 years
* Evidence of active tuberculosis or recent clinically-significant infection requiring systemic therapy.
* Evidence of active Hepatitis B, Hepatitis C, or Human Immunodeficiency virus (HIV) infection
* Have a history of brain metastasis
* Have received cancer therapies including chemotherapy, radiation, biologic, or kinase inhibitors, granulocyte-colony stimulating factor (G-CSF), or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 3 weeks prior ot the first scheduled dose of CMB305
* Female of child bearing potential who is pregnant, is planning to become pregnant, or is breast feeding; or male who is sexually active with a female of child bearing potential who is planning to become pregnant.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (27):
  - Mayo Clinic- Scottsdale, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Sarcoma Oncology Center, Santa Monica, California
  - University of Colorado Cancer Center, Boulder, Colorado
  - Yale University School of Medicine- Cancer Center, New Haven, Connecticut
  - University of Miami, Coral Gables, Florida
  - Mayo Clinic- Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center at USF, Tampa, Florida
  - Northwestern, Chicago, Illinois
  - Dana Farber Cancer Institute/Mass General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Hackensack University Medical Center, Edison, New Jersey
  - Cohen Children's Medical Center (Northwell), Astoria, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center/Seattle Cancer Care Alliance, Seattle, Washington
- Canada (2):
  - University of Alberta Hospital- Cross Cancer Institute, Edmonton
  - McGill University, Montreal East

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: CMB305 placebo control
- CMB305: CMB305: Sequentially administered LV305 [lentiviral vector encoding New York esophogeal squamous cell carcinoma-1 {NY-ESO-1} gene] and G305 [NY-ESO-1 recombinant protein plus glucopyranosyl lipid A stable emulsion {GLA-SE}]
Period: Overall Study
Arm/Group | Placebo | CMB305
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Study terminated by Sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Population: 0 participants are reported due to the risk of identification of a person.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CMB305 | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the investigator-determined date of disease progression or death, whichever comes first, using Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
Time Frame: From randomization to investigator-determined date of disease progression or death, assessed up to 24 months.
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Placebo | CMB305
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to the date of death.
Time Frame: From randomization to date of death, assessed up to 66 months.
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Placebo | CMB305
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Next Treatment (TTNT)
Description: TTNT is defined as the time from randomization to the start of post-study treatment subsequent intervention: [TTNT = start date of subsequent intervention - randomization date + 1]. Subsequent intervention includes anticancer therapy, cancer-related surgery and local regional therapy. Participants who do not start any post-study treatment intervention will be censored at their last known date of being alive.
Time Frame: From last dose of CMB305 to initiation of new therapy, assessed up to 24 months.
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Placebo | CMB305
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Distant Metastasis Free Survival (DMFS)
Description: DMFS is defined as the time from randomization to evidence of a new distant metastasis not documented at time of randomization: [DMFS = a new distant metastasis documented date - randomization date + 1]. Participants who do not have any new distant metastasis will be censored at their last tumor assessment.
Time Frame: From randomization to investigator-determined date of disease progression or death, assessed up to 24 months.
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Placebo | CMB305
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR defined by RECIST v1.1 will be summarized by the number and percent of subjects who achieve a complete response (CR) or partial response (PR) based on the investigator's assessment. ORR will be compared between treatment arms using a logistic regression.
Time Frame: From randomization to investigator-determined date of disease progression, assessed up to 24 months.
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Placebo | CMB305
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants Who Experienced a Treatment-Emergent Adverse Event (TEAE)
Description: Safety will be assessed primarily based on reported adverse events (AEs), Medical Events of Interest (MEOIs), laboratory values, and concomitant medications reported from initiation of treatment with CMB305 or placebo.
Time Frame: From randomization to investigator-determined date of disease progression or death, assessed up to approximately 2 months.
Population: All participants taking any amount of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo | CMB305
Number analyzed (Participants) | 0 | 1
Participants |  | 1

7. Secondary Outcome: Quality of Life (QoL): EuroQol 5-Dimension 5 Level (EQ-5D-5L) and EuroQol 5-Dimension Youth (EQ-5D-Y) Questionnaires
Description: QoL evaluated using the EQ-5D-5L for participants ≥18 years of age or using the EQ-5D-Y for participants 12 to <18 years of age. EQ-5D-5L descriptive system is comprised of 5 dimensions-mobility, self-care, usual activities, pain/discomfort & anxiety/depression. Each dimension has 5 levels: not at all (level 1), mild (level 2), moderate (level 3), severe (level 4), extreme/leading to incapacity (level 5), with highest level corresponding to worst outcome. Participants indicated their health state by choosing the appropriate level from each dimension. The 5 digit health states thus obtained for each dimension were then converted into a single median index value using the EQ-5D-5L crosswalk index value calculator as recommended by EuroQol group. In the EQ-VAS, participants recorded their health state on a scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: From Day 1 up to 12 months
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Placebo | CMB305
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: The number of all participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 2 months
Population: All participants taking any amount of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo | CMB305
Number analyzed (Participants) | 0 | 1
Participants |  | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 2 months
Description: 0 participants are reported due to the risk of identification of a person.
Arm/Group | Placebo | CMB305
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study was stopped early due to Sponsor decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT03520959/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT03520959/SAP_001.pdf